CLINICAL TRIAL: NCT02843464
Title: Long-term Remote Ischemic Preconditioning Improve Long-term Prognosis of Acute Myocardial Infarction Patients Without Emergency Reperfusion Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XuanwuH-RIPC2
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-07

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

ARMS (2):
- long-term RIPC group (Experimental): routine treatment + once RIPC/day for a year. Three five-minute cycles of upper limb ischaemia and three five-minute pauses using a blood pressure cuff inflated to 200 mmHg.
  Interventions: Other: reported remote ischemic preconditioning (RIPC)
- control group (No Intervention): routine treatment.

INTERVENTIONS:
Other: reported remote ischemic preconditioning (RIPC) — Three five-minute cycles of upper limb ischaemia and three five-minute pauses using a blood pressure cuff inflated to 200 mmHg.
  Arms: long-term RIPC group

SUMMARY:
Patients with acute myocardial infarction (AMI) are in critical condition especially without emergency reperfusion therapy. For example, heart failure, heart rupture, malignant arrhythmia are in high level. It was reported remote ischemic preconditioning (RIPC) may play an effective endogenous cardiac protection. This study will investigate whether long-term RIPC can improve the short-term and long-term (1 year) prognosis of AMI patients without emergency reperfusion therapy. 220 AMI patients without emergency reperfusion therapy were randomly divided into 2 groups: long-term RIPC group (once RIPC/day for a year) or control group (routine treatment). Cardiac troponin (TNI), high-sensitivity C-reactive protein (hsCRP), adenosine, vascular endothelial growth factor (VEGF), hypoxia inducible factor-1 (HIF-1), echocardiography and magnetic resonance（MR）were detected in hospital, 1 month and 1 year after discharge. Patients will be followed up by telephone at the end of one year. The major adverse cardiovascular events (MACE) include cardiovascular death, spontaneous myocardial infarction, unplanned revascularization and stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 years;
* Acute myocardial infarction (STEMI);
* Without emergency reperfusion therapy.

Exclusion Criteria:

* Age more than 80 or less than 18 years;
* Renal failure with creatinine >2 mg/dl;
* Reject taking part in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
The major adverse cardiovascular events (MACE) include cardiovascular death, spontaneous myocardial infarction, unplanned revascularization and stroke. | one year

REFERENCES:
- [Background] Tobis J. Is no-no-reflow following PCI in AMI due to distal embolization of plaque and thrombus? Catheter Cardiovasc Interv. 2013 Aug 1;82(2):210-1. doi: 10.1002/ccd.25078. No abstract available. PMID 23878032
- [Background] Crimi G, Pica S, Raineri C, Bramucci E, De Ferrari GM, Klersy C, Ferlini M, Marinoni B, Repetto A, Romeo M, Rosti V, Massa M, Raisaro A, Leonardi S, Rubartelli P, Oltrona Visconti L, Ferrario M. Remote ischemic post-conditioning of the lower limb during primary percutaneous coronary intervention safely reduces enzymatic infarct size in anterior myocardial infarction: a randomized controlled trial. JACC Cardiovasc Interv. 2013 Oct;6(10):1055-63. doi: 10.1016/j.jcin.2013.05.011. PMID 24156966
- [Background] Schmidt MR, Sloth AD, Johnsen J, Botker HE. Remote ischemic conditioning: the cardiologist's perspective. J Cardiovasc Med (Hagerstown). 2012 Nov;13(11):667-74. doi: 10.2459/JCM.0b013e328357bff2. PMID 23114270
- [Background] Szijarto A, Czigany Z, Turoczi Z, Harsanyi L. Remote ischemic perconditioning--a simple, low-risk method to decrease ischemic reperfusion injury: models, protocols and mechanistic background. A review. J Surg Res. 2012 Dec;178(2):797-806. doi: 10.1016/j.jss.2012.06.067. Epub 2012 Jul 28. PMID 22868050
- [Background] Ghaemian A, Nouraei SM, Abdollahian F, Naghshvar F, Giussani DA, Nouraei SA. Remote ischemic preconditioning in percutaneous coronary revascularization: a double-blind randomized controlled clinical trial. Asian Cardiovasc Thorac Ann. 2012 Oct;20(5):548-54. doi: 10.1177/0218492312439999. PMID 23087298
- [Background] Botker HE, Kharbanda R, Schmidt MR, Bottcher M, Kaltoft AK, Terkelsen CJ, Munk K, Andersen NH, Hansen TM, Trautner S, Lassen JF, Christiansen EH, Krusell LR, Kristensen SD, Thuesen L, Nielsen SS, Rehling M, Sorensen HT, Redington AN, Nielsen TT. Remote ischaemic conditioning before hospital admission, as a complement to angioplasty, and effect on myocardial salvage in patients with acute myocardial infarction: a randomised trial. Lancet. 2010 Feb 27;375(9716):727-34. doi: 10.1016/S0140-6736(09)62001-8. PMID 20189026
- [Background] Hausenloy DJ, Mwamure PK, Venugopal V, Harris J, Barnard M, Grundy E, Ashley E, Vichare S, Di Salvo C, Kolvekar S, Hayward M, Keogh B, MacAllister RJ, Yellon DM. Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):575-9. doi: 10.1016/S0140-6736(07)61296-3. PMID 17707752
- [Background] Shimizu M, Saxena P, Konstantinov IE, Cherepanov V, Cheung MM, Wearden P, Zhangdong H, Schmidt M, Downey GP, Redington AN. Remote ischemic preconditioning decreases adhesion and selectively modifies functional responses of human neutrophils. J Surg Res. 2010 Jan;158(1):155-61. doi: 10.1016/j.jss.2008.08.010. PMID 19540519
- [Background] Hu S, Dong HL, Li YZ, Luo ZJ, Sun L, Yang QZ, Yang LF, Xiong L. Effects of remote ischemic preconditioning on biochemical markers and neurologic outcomes in patients undergoing elective cervical decompression surgery: a prospective randomized controlled trial. J Neurosurg Anesthesiol. 2010 Jan;22(1):46-52. doi: 10.1097/ANA.0b013e3181c572bd. PMID 19996767
- [Background] Meng R, Asmaro K, Meng L, Liu Y, Ma C, Xi C, Li G, Ren C, Luo Y, Ling F, Jia J, Hua Y, Wang X, Ding Y, Lo EH, Ji X. Upper limb ischemic preconditioning prevents recurrent stroke in intracranial arterial stenosis. Neurology. 2012 Oct 30;79(18):1853-61. doi: 10.1212/WNL.0b013e318271f76a. Epub 2012 Oct 3. PMID 23035060
- [Background] D'Ascenzo F, Moretti C, Omede P, Cerrato E, Cavallero E, Er F, Presutti DG, Colombo F, Crimi G, Conrotto F, Dinicolantonio JJ, Chen S, Prasad A, Biondi Zoccai G, Gaita F. Cardiac remote ischaemic preconditioning reduces periprocedural myocardial infarction for patients undergoing percutaneous coronary interventions: a meta-analysis of randomised clinical trials. EuroIntervention. 2014;9(12):1463-71. doi: 10.4244/EIJV9I12A244. PMID 24755386
- [Background] Liu Z, Wang YL, Hua Q, Chu YY, Ji XM. Late remote ischemic preconditioning provides benefit to patients undergoing elective percutaneous coronary intervention. Cell Biochem Biophys. 2014 Sep;70(1):437-42. doi: 10.1007/s12013-014-9936-1. PMID 25015066